CLINICAL TRIAL: NCT05403385
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study Evaluating Efficacy and Safety of Inupadenant in Combination With Carboplatin and Pemetrexed in Adults With Nonsquamous Non-small Cell Lung Cancer Who Have Progressed on Immunotherapy
Brief Title: Study of Inupadenant (EOS100850) With Chemotherapy as Second Line Treatment for Nonsquamous Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: iTeos Therapeutics (Industry)
Collaborators: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A2A-005; 2024-515393-27-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-18; First posted 2022-06-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer; Locally Advanced NSCLC - Non-Small Cell Lung Cancer
Keywords: non-squamous NSCLC; second line; 2L; adenosine; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Part 1 sequential dose escalation. Part 2 randomized double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple masking : The dose-finding part (Part 1) of this study is open-label whereas the randomized part (Part 2) is double-blinded. Therefore, for Part 2, the subject, the Investigator and Sponsor personnel or delegate(s) who are involved in the treatment administration or clinical evaluation of the subjects will be unaware of the group assignments. The chemotherapy agents administered during Part 2 will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1, open label (Experimental): Inupadenant will be given at one or more dose levels to determine the recommended Phase 2 dose (RP2D).
  Interventions: Drug: inupadenant; Drug: Carboplatin; Drug: Pemetrexed
- Part 2, active treatment (Experimental): Treatment with inupadenant combined with carboplatin and pemetrexed
  Interventions: Drug: inupadenant; Drug: Carboplatin; Drug: Pemetrexed
- Part 2, placebo (Placebo Comparator): Treatment with matched placebo combined with carboplatin and pemetrexed
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: inupadenant — Adenosine 2a receptor antagonist
  Other Names: EOS100850
  Arms: Part 1, open label; Part 2, active treatment
Drug: Placebo — matched placebo capsule to inupadenant
  Arms: Part 2, placebo
Drug: Carboplatin — standard of care chemotherapeutic, alkylating agent
Drug: Pemetrexed — standard of care chemotherapeutic, anti-metabolite
  Other Names: Alimta

SUMMARY:
The study will first determine the optimal dose of inupadenant to be given in combination with carboplatin and pemetrexed to patients that progressed after receiving first line anti-PD(L)1 treatment for locally advanced or metastatic non-small cell lung cancer. The efficacy and safety of the combination is then compared to standard of care carboplatin and pemetrexed in the same populations.

DETAILED DESCRIPTION:
The study is composed of two parts. Part 1 follows an open-label, dose-finding design where individual cohorts are treated with various dose levels of inupadenant combined with standard of care dosing of carboplatin and pemetrexed. The recommended phase 2 dose is determined prior to initiation of Part 2 which then compares inupadenant to placebo with both arms treated in combination with standard of care carboplatin and pemetrexed.

Participants in both parts are enrolled from two populations of patients with nonsquamous NSCLC that have progressed after first line treatment as follows: non-resectable patients treated with chemoradiotherapy followed by anti-PD-(L)1 or metastatic patients treated with anti-PD-(L)1 therapy without chemotherapy.

Imaging, safety and PRO assessments are performed during the treatment and follow-up phase as well as pharmacokinetic and other exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic (Stage IV) or locally advanced, unresectable (Stage III) NSCLC of nonsquamous pathology
* Measurable disease as defined by RECIST v1.1
* PD-L1 expression status available at or after the time of diagnosis. All levels of expression are eligible.
* Existing biopsy taken within 4 years prior to entering trial or provide fresh biopsy where safe and feasible
* At least 12 weeks of treatment with only 1 anti-PD-(L)1 agent (mono or with IO combo) in the metastatic setting, OR at least 12 weeks of anti-PD-(L)1 agent (mono or with IO combo) following CRT in the unresectable, Stage III setting
* ECOG performance status of 0 to 1.

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases or leptomeningeal disease.
* EGFR, ALK, or ROS1 mutation.
* Autoimmune disease requiring systemic treatment or immunodeficiency requiring concurrent use of systemic immunosuppressants or corticosteroids
* Hepatitis B or C infection unless adequately treated with no detectable viral load; Human immunodeficiency virus (HIV) unless well-controlled disease on therapy.
* History of life-threatening toxicity related to prior immune therapy
* Uncontrolled or significant cardiovascular disease
* Pregnant or breast-feeding
* Lack of agreement to use highly effective method of contraception during treatment and for 6 months after the last administration of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Dose-finding to determine recommended Phase 2 dose | At the end of Cycle 1 (each cycle is 21 days)
  Incidence of dose-limiting toxicities
Incidence of treatment-emergent adverse events [Safety and Tolerability] | Duration of intervention (up to 24 months) plus 30 days follow-up or up to database lock
  Incidence of adverse events (AEs), serious adverse events, AEs leading to discontinuation, deaths, and clinically significant laboratory abnormalities.
Progression-free survival [Efficacy] | From randomization to first-documented radiological progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  Time from first dose to the date of first documented radiologic progression per RECIST v1.1 or time of death, whichever comes first

SECONDARY OUTCOMES:
Overall Response Rate [Efficacy] | From randomization to first-documented radiological improvement, if applicable, assessed up to 24 months or up to database lock.
  Proportion of participants with a best overall response of complete (CR) or partial (PR) response as assessed by RECIST v1.1
Duration of Response [Efficacy] | From first-documented CR or PR to first radiological progression or date of death, whichever comes first, assessed up to 24 months or up to database lock.
  Time from first CR or PR to first documented progression or death from any cause, per RECIST v1.1
Percent Change in Tumor Size [Efficacy] | From randomization to the documented radiological assessment with the smallest tumor size sum, assessed up to 24 months or up to database lock.
  Change in sum of size of target tumors from baseline, per RECIST v1.1
Disease Control Rate [Efficacy] | From randomization to second-documented radiological CR, PR or SD, if applicable, assessed up to 24 months or up to database lock.
  Proportion of participants with CR, PR, or stable disease (SD) sustained over at least 2 consecutive tumor assessments, per RECIST v1.1
Overall Survival [Efficacy] | From randomization to death due to any cause, assessed up to 24 months or up to database lock.
  Time from randomization to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Belgium SA
Locations (21):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Lucas, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Delta, Roeselare
- William Osler Health System, Brampton, Ontario, Canada
- Vseobecna Fakultni Nemocnice, Prague, Czechia
- France (3):
  - CHU de Caen, Caen
  - Hopital de la Timone Centre d'Essais Précoces en Cancérologie de Marseille (CEPCM), Marseille
  - CHU Nantes, Nantes
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan
  - Gruppo Humanitas - Istituto Clinico Humanitas, Rozzano
- Spain (8):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario de Navarra (CHN), Pamplona, Pamplona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Valencia
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Infanta Cristina (Hospital Universitario de Badajoz), Badajoz
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Althaia Hospital, Manresa
  - Complejo Hospitalario Universitario de Ourense, Ourense
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No